CLINICAL TRIAL: NCT07114315
Title: A Phase II Clinical Study of AK130 in Combination With AK112 for the Treatment of Advanced Pancreatic Cancer
Brief Title: A Study of AK130 in Combination With AK112 for the Treatment of Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK130-202
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 in combination with AK130 (Experimental)
  Interventions: Drug: AK112; Drug: AK130
- AK112 (Experimental)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — Following a predefined dose and date.
Drug: AK130 — Following a predefined dose and date.
  Arms: AK112 in combination with AK130

SUMMARY:
This is an open-label, multi-center phase II clinical study consisting of two parts:

Part I: To evaluate the safety and efficacy of AK130 combined with AK112 in advanced pancreatic cancer.

Part II: To evaluate the safety and efficacy of AK112, either as monotherapy or in combination with AK130, in advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent.
2. Have a life expectancy of at least 3 months.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Subjects with histologically or cytologically confirmed advanced/metastatic pancreatic ductal adenocarcinoma (PDAC), who have progressed on ≤2 prior lines of systemic therapy.
5. According to RECIST v1.1, there is at least one measurable lesion.
6. Has adequate organ function.
7. All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 90 days after the last dose of study treatment.
8. Able to to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

1. Except for PDAC, the subjects had other malignant tumors within the 5 years prior to enrollment.
2. There is central nervous system (CNS) metastasis, spinal cord compression, or meningeal metastasis.
3. There are pleural effusion, pericardial effusion, or ascites with clinical symptoms or requiring repeated drainage.
4. Prior systemic therapy with either TGF-β inhibitors or anti-angiogenic agents.
5. There is a history of non infectious pneumonia that requires systemic glucocorticoid treatment.
6. History of severe bleeding tendency or coagulation dysfunction.
7. Previous history of myocarditis, cardiomyopathy, and malignant arrhythmia.
8. Pregnant or lactating female subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | From the time of informed consent signed through 30 days after the last dose of study drug or starting new anti-cancer therapy.
  AE refers to any untoward medical occurrence or deterioration of existing medical event after the subject signed the ICF, whether or not considered related to the study treatment.
Objective Response Rate (ORR) | Through study completion, an average of 2 years
  ORR is defined as the proportion of subjects with BOR response of CR or PR (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
Disease control rate (DCR) | Through study completion, an average of 2 years
  DCR is defined as the proportion of subjects with response of CR, PR and SD (based on RECIST Version 1.1).
Duration of Response (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  The time from first documented evidence of CR or PR until time of first documented disease progression.
Time to response (TTR) | From date of randomization until the date of first documented response, assessed up to 24 months.
  Time between date of start of treatment until first documented response (CR or PR).
Progression Free Survival (PFS) | Through study completion, an average of 2 years.
  PFS is defined as the interval between first dose and the earliest date of disease progression or death due to any cause.
Overall survival (OS) | Through study completion, an average of 2 years.
  OS is defined as the time from first dose until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No